CLINICAL TRIAL: NCT00546780
Title: Phase 3 Randomized, Open-Label Clinical Trial of Tanespimycin (KOS-953) Plus Bortezomib Compared to Bortezomib Alone in Patients With Multiple Myeloma in First Relapse
Brief Title: A Study of Tanespimycin (KOS-953) in Patients With Multiple Myeloma in First Relapse
Acronym: BMS TIME-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA200-004; KAG-301
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Heat Shock Protein 90; Hsp90; KOS-953; 17-AAG; bortezomib; first relapse; tanespimycin; TIME-1
MeSH Terms: conditions — Multiple Myeloma | interventions — tanespimycin; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Tanespimycin + Bortezomib
  Interventions: Drug: Tanespimycin; Drug: Bortezomib
- Arm B (Active Comparator): Bortezomib
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Tanespimycin — Solution, IV, 340mg/m2, twice weekly for 2 weeks (3 week cycle), 60 minutes infusion
  Other Names: BMS-722782
  Arms: Arm A
Drug: Bortezomib — Solution, IV, 1.3 mg/m2, twice weekly for 2 weeks (3 weeks cycle), 3-5 minute bolus

SUMMARY:
This is a phase 3, open label trial for patients with multiple myeloma in first relapse. Trial will compare tanespimycin (KOS-953), in combination with a fixed dose of bortezomib versus bortezomib alone.

DETAILED DESCRIPTION:
Phase 3 combination study comparing tanespimycin (KOS-953) plus bortezomib to bortezomib alone in patients with multiple myeloma in first relapse after failure of previous anti-cancer therapy and/or bone marrow transplantation. Primary objective is to compare the progression-free survival (PFS) associated with the use of tanespimycin (KOS-953) in combination with bortezomib versus that associated with administration of bortezomib alone.

ELIGIBILITY:
Inclusion Criteria:

* Good Performance Status
* Documented evidence of multiple myeloma
* Documented progression of disease after initial response to one line of therapy
* Measurable disease (serum M-protein >.5g/dl or > 200 mg urinary M protein excretion)

Exclusion Criteria:

* Prior treatment with a heat shock 90 inhibitor or an investigational proteasome inhibitor
* Known active infections of HAV, HBV, HCV, or HIV
* Administration of chemotherapy, radiation therapy, or immune therapy within 21 days prior to randomization.
* Acute diffuse infiltrate pulmonary disease or pericardial dise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6-24 months

SECONDARY OUTCOMES:
Overall survival in each arm of the study | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (18):
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - Moores Ucsd Cancer Center, La Jolla, California
  - University Of California Medical Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - University Of Kansas Medical Center, Westwood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System Irb, Detroit, Michigan
  - Capitol Comprehensive Cancer Care Center, Jefferson City, Missouri
  - Columbia University Medical Center (Cumc), New York, New York
  - Wake Forest Univ Health Sciences, Winston-Salem, North Carolina
  - Kaiser Permanente Oncology/Hematology, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Local Institution, Edmonton, Alberta, Canada

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx